CLINICAL TRIAL: NCT03761953
Title: A Pilot Proof of Concept Single-Center Study of the Use of Oritavancin in Systemic Staphylococcus Aureus Infections in Patients With Opioid Use Disorder
Brief Title: Oritavancin for Staphylococcus Aureus Infections in Opioid Users
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: COVID 19 pandemic
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 831334
Record Dates: First submitted 2018-11-09; First posted 2018-12-03 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2022-03

CONDITIONS: Staphylococcus Aureus Bacteremia; Staphylococcus Aureus Endocarditis
MeSH Terms: interventions — oritavancin

STUDY DESIGN:
Intervention Model Description: This will be a pilot single-arm study consisting of 15 patients evaluating the use of oritavancin in the final consolidation phase (last two weeks of treatment) of systemic infections with Staphylococcus aureus (S. aureus) in opioid users.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Oritavancin (Experimental): Single IV infusion of 1200mg of oritavancin
  Interventions: Drug: Oritavancin Injection

INTERVENTIONS:
Drug: Oritavancin Injection — single 1200mg infusion of IV oritavancin.

SUMMARY:
This will be a pilot single-arm study consisting of 15 participants evaluating the use of oritavancin in the final consolidation phase (last two weeks of treatment) of systemic infections with Staphylococcus aureus (S. aureus) in opioid users.

The purpose of this pilot proposal is to collect information for a subsequent large, randomized intervention. Primary endpoints will be 1) Safety and tolerability, and 2) Duration of hospitalization and rate of recurrence.

DETAILED DESCRIPTION:
This will be an early phase, single center, open label pilot study of 15 participants designed to evaluate the effects of oritavancin in patients with Opioid Use Disorder and/or Intravenous Drug Use and systemic S. aureus infections. In this study systemic infections refers to bacteremia or Infectious Endocarditis. Participants who meet inclusion and exclusion criteria will receive a single 1200mg infusion of oritavancin to complete 4 weeks of antibiotic therapy (including the inpatient phase) for isolated bacteremia and 6 weeks for IE. Participants will be evaluated weekly until completion of treatment and then at week 4 and week 6 after the infusion of oritavancin. Participants will have blood drawn at each visit to monitor for toxicity and pharmacokinetics and will be evaluated clinically and by culture for the presence of relapse of the infection. At the last visit, participants will have an echocardiogram.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age and older
* Systemic infection with S. aureus
* Afebrile for >48 hours
* Negative blood cultures for at least 48 hours
* Absolute neutrophil count (ANC) equal or greater 750/mm3
* Hemoglobin > 9.0 g/dL
* Platelet count equal or > 50,000/mm3
* Creatinine < 2.0 x ULN
* AST ; ALT, and alkaline phosphatase < 2.0 x ULN
* Willing to use a medically accepted method of contraception

Exclusion Criteria:

* Require valve replacement surgery
* Have prosthetic material in body (This includes prosthetic heart valves and/or prosthetic joints)
* Septic emboli to central nervous system or lungs
* Breast feeding during entire participation
* Pregnant
* Polymicrobial infection
* Require anticoagulation
* Allergy to vancomycin or oritavancin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2022-03-24 (Actual); Study Completion 2022-03-24 (Actual)

PRIMARY OUTCOMES:
Frequency of grade 3 or 4 systemic (i.e., not a local reaction) adverse events associated with the administration of oritavancin | 6 weeks
  Safety
Frequency of relapse of infection | 6 weeks
  Efficacy

SECONDARY OUTCOMES:
Duration of hospitalization | 6 weeks
  Duration of hospitalization
Relapse of systemic S. aureus infections | 6 weeks
  Relapse of systemic S. aureus infections. Relapse will be defined as an isolation of the same S. aureus strain in subsequent cultures
Pharmacokinetic parameters of oritavancin: Cmin (μg/ml) | 6 weeks
  Cmin (μg/ml) at week 1, 2, 4 and 6 after the administration of oritavancin
Patient satisfaction when using oritavancin measured using the Patient Satisfaction Questionnaire Short Form (PSQ-18) | 6 weeks
  Patient satisfaction will be measured using The Patient Satisfaction Questionnaire Short Form (PSQ-18)

CONTACTS AND LOCATIONS:
Overall Officials: Pablo Tebas, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- Clinical Trials Unit. University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No